CLINICAL TRIAL: NCT04939519
Title: SCALE-UP Utah: Community-Academic Partnership to Address COVID-19 Among Utah Community Health Centers
Brief Title: SCALE-UP Utah: Community-Academic Partnership to Address COVID-19 Vaccination Rates Among Utah Community Health Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Association for Utah Community Health (Other); Utah Department of Health (Other); National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, David Wetter, Director, Center for Health Outcomes and Population Equity, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 00136001_2; 3UL1TR002538-03S2 (NIH)
Record Dates: First submitted 2021-04-07; First posted 2021-06-25 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Covid19
Keywords: COVID19; Community Health; Health Information Technology; Population Health; Patient engagement; Rural; Scale up; Screening; vaccinations; Text messaging; Underserved population; Uninsured; Utah; Uptake; Population Health Tool
MeSH Terms: conditions — COVID-19; Patient Participation | interventions — Patient Navigation

STUDY DESIGN:
Intervention Model Description: Patient-level, two-arm randomized design for the Population Health Management interventions, TM or TM+PN.
Who Masked: Participant
Masking Description: Patients will not know if they are in the TM or TM+PN intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text-Messaging (TM) (Active Comparator): Population health management intervention that analyzes electronic health record data to automatically identify participants who are eligible for the COVID-19 vaccine and proactively reach those participants for vaccine scheduling. This is a bi-directional text messaging system.
  Interventions: Behavioral: Text-Messaging (TM)
- Text-Messaging plus Patient Navigation (Active Comparator): Population health management intervention that includes the same bi-directional text-messaging system as Arm 1 (the text messaging condition) with the addition of patient navigation. Patient navigation includes real-time assistance from a community health worker to address barriers, provide motivation, and assist with logistics of COIVD vaccination.
  Interventions: Behavioral: Text-Messaging (TM); Behavioral: Patient Navigation (PN)

INTERVENTIONS:
Behavioral: Text-Messaging (TM) — Participants in the TM condition will receive HIPAA-compliant bidirectional text messages. These texts will include a brief message alerting patients that they are eligible to receive the vaccine and asking participants if they would like to schedule a vaccine. Participants who reply "yes" will receive an additional message with information about how and where to register for the vaccine. This information will vary depending on local availability. Participants who reply "no" will receive a text requesting they contact their local clinic when they decide to receive the vaccine.
Behavioral: Patient Navigation (PN) — Participants in the PN condition will receive a message alerting them that a Community Health Worker will contact them to assist with the process of scheduling a vaccine. At this time the participant has the option to opt-out of this follow up phone call. The patient navigation from the Community Health Worker includes practical advice in addressing barriers to vaccination such as logistics and transportation, as well as fear, skepticism, and hesitancy.
  Arms: Text-Messaging plus Patient Navigation

SUMMARY:
SCALE-UP Utah is a community-academic partnership to address COVID-19 among Utah community health centers. The long-term objective of the project is to increase the reach, acceptance, and uptake of COVID-19 vaccines among Utah's Community Health Center patient population. The study will compare two practical, feasible, scalable interventions to increase COVID-19 vaccine uptake in Utah Community Health Centers:

1. Text Messaging (TM): population health management (PHM) intervention that analyzes EHR data to automatically identify patients eligible for COVID-19 vaccination and uses bi-directional text messaging to help connect patients to a vaccination site;
2. Patient Navigation (PN): PHM intervention to increase vaccination uptake among eligible patients (identified via TM) using patient navigation (e.g., motivating patients, addressing logistics and barriers).

The project will employ a rapid cycle research approach in which interventions are tested on a small scale, using short time frames (e.g., <1 month) and cyclical evaluation cycles.This process involves implementing intervention messages with a small number of clinics or patients, evaluating the outcomes, and either adapting the intervention messages based on findings (and retesting) or disseminating effective approaches to additional clinics or patients. A critical feature of these cycles is the ability to quickly test and refine messages in a limited setting before broader implementation. Throughout the study, intervention messages were updated or adapted in response to evolving public health guidelines, testing procedures, and policy recommendations (e.g., priority populations by age group or geographic area, as advised by the Utah Department of Health and Human Services and relevant federal agencies). However, these updates did not alter the fundamental structure of the intervention arms. Participants were randomized to one of two main conditions-Text Messaging (TM) or Text Messaging plus Patient Navigation (TM+PN)-and all participants within a given arm received interventions aligned with their assigned condition. Adaptations occurred within the content and timing of messages or navigation support, but the core components of the interventions remained consistent across participants within each arm. These adaptations were tracked and incorporated into implementation logs but did not constitute distinct intervention arms or conditions.

The specific aims are to:

1. Implement and evaluate PHM interventions for increasing the uptake of COVID-19 vaccinations among CHC patients across Utah. Our primary outcome, Uptake-Eligible, is defined as the proportion of patients who receive a COVID-19 vaccination out of those who meet eligibility criteria for vaccination. Our study hypothesis is that patients in the TM+PN cohort will have higher rates of uptake-eligible than those in the TM cohort.
2. Examine implementation effectiveness outcomes, as well as characteristics of both clinics and patients that may influence intervention effects and implementation outcomes.

DETAILED DESCRIPTION:
SCALE-UP Utah is a patient-level intervention involving 12 Community Health Centers (39 individual clinics) across Utah. The study is designed to utilize Community Health Center patient records to proactively reach patients for COVID-19 vaccinations. This intervention includes a randomization component between two interventions, text messaging (TM) or text messaging with patient navigation (TM+PN). These two intervention paths are occurring simultaneously within the same clinics.

Text messaging (TM) and text messaging with patient navigation (TM+PN)

Overview:

Participants in the TM condition will receive HIPAA-compliant bidirectional text messages. These texts will include a brief message alerting patients that they are eligible to receive the vaccine and asking participants if they would like to schedule a vaccine. Participants who reply "yes" will receive an additional message with information about how and where to register for the vaccine. This information will vary depending on local availability. Participants who reply "no" will receive a text requesting they contact their local clinic when they decide to receive the vaccine.

Participants in the TM+PN condition will receive the same text message as the participants in the TM condition. Texts will include a brief message alerting patients that they are eligible to receive the vaccine and asking participants if they would like to schedule a vaccine. Participants who reply "yes" will receive the same information about how and where to receive a vaccine however, they will also receive a message alerting them that a Community Health Worker will contact them to assist with this process, in case they need that. At this time the participant has the option to opt-out of this follow up phone call. The patient navigation from the Community Health Worker includes practical advice in addressing barriers to vaccination such as logistics and transportation, as well as fear, skepticism, and hesitancy.

Step One: Primary Data Extraction To identify the cohort for the TM and TM+PN interventions, a subset of EHR data will be manually extracted from the Community Health Centers as text files generated by EHR reports. The first set of EHR reports will contain all patients seen at each of the Community Health Centers in the last 3 years. Subsequent reports will be obtained weekly, including all encounters in the previous week. Data fields will include risk factors such as age, gender, body mass index, encounter diagnoses for medical co-morbidities, patient demographics (e.g., zip code, insurance status, preferred language, race/ethnicity); as well as cellphone number for text messaging and patient navigation.

Step Two: Randomization & Cohort Selection. Once the data are securely housed, all patients will be assigned to either the TM or TM+PN arm of the intervention. This assignment will remain consistent throughout the study. Cohort selection for the text messages will be based on EHR data considering factors such as age, race/ethnicity, language, relevant medical comorbidities, and residence in low-vaccination areas. These selection criteria are consistent with recommendations from Utah Department of Health and the Centers for Disease Control and Prevention.

Step Three: Implementation. SCALE-UP Utah will send HIPPA-compliant bidirectional texts, which is a communication method routinely used by the Community Health Centers, to patients who are eligible for COVID-19 vaccination. Text messages will be designed by the research team and sent using a HIPPA compliant text messaging service. The text messaging service will retrieve the patient cohort from the study database to send the texts to the patients. The text messages will appear to the patients as having originated from their Community Health Center. As part of their general Community Health Center care, patients have agreed to be contacted by their Community Health Center and text message communication is one of those established contact methods. Text messages will be repeated bi-weekly to continuously prompt vaccination update. This process will repeat until the participant indicates that they have either scheduled or received their vaccination. Every text message will include the option to reply STOP to opt-out of receiving text messages at any time.

ELIGIBILITY:
Inclusion Criteria:

* current patient of a participating community health center
* have a working cellphone,
* have phone number listed in existing electronic medical record at their participating clinic
* speak English or Spanish.

Exclusion Criteria:

* Minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65300 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wetter, MS, PhD, Principal Investigator — University of Utah; Rachel Hess, MD, MS, Principal Investigator — University of Utah; Guilherme Del Fiol, MD, PhD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute/ University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Text-Messaging (TM) | Text-Messaging Plus Patient Navigation
Started | 32594 | 32706
Completed | 32594 | 32706
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text-Messaging (TM) | Text-Messaging Plus Patient Navigation | Total
Number analyzed (Participants) | 32594 | 32706 | 65300
Age, Customized [Count of Participants; unit: Participants]
  18-29 years old | 9210 | 9096 | 18306
  30-64 years old | 19902 | 20033 | 39935
  65 and older | 3482 | 3577 | 7059
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 17535 | 17376 | 34911
  Male | 13387 | 13687 | 27074
  Other or unknown | 1672 | 1643 | 3315
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12792 | 12820 | 25612
  Not Hispanic or Latino | 16201 | 16324 | 32525
  Unknown or Not Reported | 3601 | 3562 | 7163
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native White | 728 | 763 | 1491
  Asian | 206 | 241 | 447
  Black or African American | 380 | 330 | 710
  Native Hawaiian or Pacific Islander | 226 | 217 | 443
  More than one race | 444 | 445 | 889
  Other Race | 3602 | 3561 | 7163
  White | 21888 | 22002 | 43890
  Unknown or Not Reported | 5120 | 5147 | 10267

OUTCOME MEASURES:

1. Primary Outcome: Uptake-Total
Description: Proportion of patients who receive a COVID-19 vaccine out of the total patient population
Time Frame: 12 months
Population: Proportion of patients who receive a COVID-19 vaccine out of the total patient population
Measure: Count of Participants; unit: Participants
Arm/Group | Text-Messaging (TM) | Text-Messaging Plus Patient Navigation
Number analyzed (Participants) | 32594 | 32706
Participants | 14308 | 14381

2. Secondary Outcome: Reach-TM Engage
Description: Proportion of patients that respond to the Text Messaging intervention
Time Frame: 12 months
Population: Proportion of patients that respond to the Text Messaging intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Text-Messaging (TM) | Text-Messaging Plus Patient Navigation
Number analyzed (Participants) | 32594 | 32706
Participants | 5538 | 5587

3. Secondary Outcome: Reach-PN Engage- Logistics Assistance
Description: Proportion of patients offered Logistics Assistance Patient Navigator (PN-LA) that talk to a PN
Time Frame: 12 months
Population: Proportion of patients offered Logistics Assistance Patient Navigator (PN-LA) that talk to a PN
Measure: Count of Participants; unit: Participants
Arm/Group | Text-Messaging (TM) | Text-Messaging Plus Patient Navigation
Number analyzed (Participants) | 0 | 1469
Participants | 0 | 592

4. Secondary Outcome: Reach-PN Engage- Requested Navigation
Description: Proportion of patients offered Requested Navigation Patient Navigator (PN-RN) that talk to a PN
Time Frame: 12 months
Population: Proportion of patients offered Requested Navigation Patient Navigator (PN-RN) that talk to a PN
Measure: Count of Participants; unit: Participants
Arm/Group | Text-Messaging (TM) | Text-Messaging Plus Patient Navigation
Number analyzed (Participants) | 0 | 175
Participants | 0 | 122

ADVERSE EVENTS:
Time Frame: This project used a non-systematic assessment method to evaluate adverse events. Although adverse events were not routinely assessed, data on adverse events were collected for up to 23 months after a participant's enrollment in the project.
Description: Adapted intervention refers to the adaptation of messages, not interventions. Throughout the study, intervention messages were updated or adapted in response to evolving public health guidelines, testing procedures, and policy recommendations These updates did not alter the fundamental structure of the intervention arms and did not constitute distinct intervention arms.
Arm/Group | Text-Messaging (TM) | Text-Messaging Plus Patient Navigation
All-Cause Mortality (participants affected / at risk) | 0/32594 | 0/32706
Serious Adverse Events (participants affected / at risk) | 0/32594 | 0/32706
Other Adverse Events (participants affected / at risk) | 0/32594 | 0/32706

LIMITATIONS AND CAVEATS:
During the analysis portion of this project, the investigators decided that the original primary outcome and a secondary outcome were duplicative due to the eventual widespread availability of the COVID-19 Vaccine. Therefore, the investigators decided to delete the primary outcome and keep the secondary outcome as the primary. Study protocol and Statistical Analytic plan were amended to reflect the changes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/19/NCT04939519/Prot_000.pdf